CLINICAL TRIAL: NCT05830435
Title: Trier Social Stress Test in Virtual Reality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: University of Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: TSST-VR
Record Dates: First submitted 2023-03-13; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Stress, Psychological; Stress, Physiological
MeSH Terms: conditions — Stress, Psychological | interventions — Psychological Tests

STUDY DESIGN:
Intervention Model Description: In this study, a three-arm single blind randomized placebo-controlled trial will be conducted. The following conditions will be set up.
  1. TSST-VR Friendly (control)
  2. TSST-VR-Neutral
  3. TSST-VR-Unfriendly Participants will be divided into three groups by means of block randomization
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TSST VR Friendly (Active Comparator)
  Interventions: Behavioral: Trier social stress test
- TSST VR Neutral (Experimental)
  Interventions: Behavioral: Trier social stress test
- TSST VR Unfriendly (Experimental)
  Interventions: Behavioral: Trier social stress test

INTERVENTIONS:
Behavioral: Trier social stress test — TSST-VR-friendly: The assistant behind the desk asks the participant to prepare a small talk on their favourite holiday within 5 minutes. Then the participant is asked to tell about his holiday for 5 minutes. Then the participant is asked to do a simple math task: adding the number 5 to 0 for 5 minutes. The research assistant gives friendly gestures and verbal encouragements. TSST-VR-neutral: The assistant asks the participant to prepare a speech for a job interview in the upcoming 5 minutes. Then the participant is asked to deliver the speech for 5 minutes in front of two panelists and camera. Then the participant is asked to do a math task, subtracting the number 13 from 1022 for 5 minutes. During the performance the two panellist have neutral gestures and give neutral verbal instructions. TSST-VR unfriendly: The procedure of the TSST-VR unfriendly is the same as the neutral TSST-VR, with the addition that the two panellist give unfriendly gestures such as tapping on the table.

SUMMARY:
Background The Trier Social Stress Test (TSST) is a valid and gold standard way for inducing psychosocial stress and is widely used in research and diagnostics. One of the downsides of the TSST is the difficulty to maintain the same experimental conditions repeatedly. A TSST in virtual reality (TSST-VR) is constant and requires far less time and personnel. Our TSST-VR version consist of three stress levels (no stress, moderate stress, high stress), a novelty in this field.

Aim The aim is to investigate whether there is a statistically significantly greater increase directly after the TSST-VR in psychological and physiological stress parameters in the moderate and high stress levels compared to the no stress condition (control).

Method A randomized controlled trial is conducted in healthy adults, with the three stress levels as conditions. Cortisol and questionnaires on anxiety and physical arousal are measured at baseline, during and after the TSST. Heart rate is measured continuously and adverse events are monitored.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants, not having a psychiatric diagnosis in the last three years or currently having an endocrine disorders
* Aged between 18 and 65 years
* Good understanding of the Dutch language
* Normal or corrected-to-normal vision and hearing

Exclusion Criteria:

* History of photosensitive epilepsy
* Hearing loss
* Pregnant woman
* Women who breastfeed
* Taking heart rate altering medication such as beta-blockers.

Pregnant woman and woman who breastfeed are excluded because they have a different hormone levels which can intervene with the stress reaction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of levels of physical stress, HRV | continuously during the whole procedure, in total 75 minuten
  Change from baseline to 75 min

SECONDARY OUTCOMES:
Change of levels of psychological stress, state anxiety inventory STAI | After 20 minutes waiting period, after the stress test (+15min), after another 20min waiting period, and after another 20min waiting period.
  Change from baseline to the last waiting period. 6 questions each scoring 1-4, with a total score of 24. A higher score indicates for more stress and anxiety.
Social phobia | Baseline
  Social phobia scores measured by the Social Phobia Inventory
Sociodemographics | baseline
  Age, gender, work
Speech fluency | during the speech and math task, 10 minutes in total
  Speech fluency as recorded during the speech and math task
Change of levels of physical stress, cortisol | After 20 minutes waiting period, after the stress test (+15min), after another 20min waiting period, and after another 20min waiting period.
  Change from baseline to the last waiting period
Change of levels of physical stress, Skin conductance | continuously during the whole procedure, in total 75 minuten
  Galvanic Skin Conductance

CONTACTS AND LOCATIONS:
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirschbaum C, Pirke KM, Hellhammer DH. The 'Trier Social Stress Test'--a tool for investigating psychobiological stress responses in a laboratory setting. Neuropsychobiology. 1993;28(1-2):76-81. doi: 10.1159/000119004. PMID 8255414
- [Background] Helminen EC, Morton ML, Wang Q, Felver JC. Stress Reactivity to the Trier Social Stress Test in Traditional and Virtual Environments: A Meta-Analytic Comparison. Psychosom Med. 2021 Apr 1;83(3):200-211. doi: 10.1097/PSY.0000000000000918. PMID 33534392